CLINICAL TRIAL: NCT06240845
Title: Effect of High Versus Low-level Laser Therapy in Patients of Lumber Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0239
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Lumbar Radiculopathy
Keywords: HLLT, Laser therapy , LLLT, Lumber radiculopathy, Sciatica
MeSH Terms: conditions — Radiculopathy; Sciatica | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Level Laser Therapy (Experimental): This group received High-level laser therapy along with conventional physiotherapy treatment 3 times per week for 6 weeks.
  Interventions: Other: High-level laser therapy
- Low Level Laser Therapy (Experimental): This group received Low-level laser therapy along with conventional physiotherapy treatment 3 times per week for 6 weeks.
  Interventions: Other: Low-level laser therapy

INTERVENTIONS:
Other: High-level laser therapy — This group received High-level laser therapy along with conventional physiotherapy treatment 3 times per week for 6 weeks.
  Arms: High Level Laser Therapy
Other: Low-level laser therapy — This group received Low-level laser therapy along with conventional physiotherapy treatment 3 times per week for 6 weeks.
  Arms: Low Level Laser Therapy

SUMMARY:
To Compare the effects of high-level laser therapy (HLLT) and low-level laser therapy (LLLT) on pain in patients with lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders male and female will be included.
* Patients aged 40-65 years will be included.
* Patients with a diagnosis of lumbar radiculopathy confirmed by clinical evaluation by a physician or physiotherapist.
* Patients with a history of radicular leg pain and/or numbness or tingling sensation in the leg.
* a positive score on the Straight Leg Raise (pain between 35 degrees and 75 degrees), pain limiting functional ability, and scores at least 3/10 on the VAS, restricted lumbar range of motion - 25% flexion, 20% extension.
* Patients who have not received any form of treatment for lumbar radiculopathy within the past 3 months

Exclusion Criteria:

* Patients with a history of spinal surgery in the last 2 years or spinal deformity.
* Patients with a history of fracture or dislocation of the lumbar spine.
* Patients with a diagnosis of any other neurological disorder or neuropathy.
* Patients who are pregnant or breastfeeding.
* Patients with any other medical condition that may interfere i.e. inflammatory rheumatic disease, cardiac pacemaker, continuing that may interfere with the study outcomes or put them at risk with the study outcomes or put them at risk.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Pain Level | 6 weeks
  Visual Analogue scale
Rang of motion | 6 weeks
  Straight Leg Raise
Level of Disability | 6 weeks
  Oswestry Disability Index (ODI)
To measure Quality of Life | 6 weeks
  Health Questionnaire (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (2):
- Pakistan (2):
  - Faiq Medical Complex, Faisalābad, Punjab Province
  - Independent University Hospital, Faisalābad, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolu E, Buyukavci R, Akturk S, Eren F, Ersoy Y. Comparison of high-intensity laser therapy and combination of transcutaneous nerve stimulation and ultrasound treatment in patients with chronic lumbar radiculopathy: A randomized single-blind study. Pak J Med Sci. 2018 May-Jun;34(3):530-534. doi: 10.12669/pjms.343.14345. PMID 30034410
- [Background] Ince S, Eyvaz N, Dundar U, Toktas H, Yesil H, Eroglu S, Adar S. Clinical Efficiency of High-Intensity Laser Therapy in Patients With Cervical Radiculopathy: A 12-Week Follow-up, Randomized, Placebo-Controlled Trial. Am J Phys Med Rehabil. 2024 Jan 1;103(1):3-12. doi: 10.1097/PHM.0000000000002275. Epub 2023 May 1. PMID 37204965
- [Background] Konstantinovic LM, Cutovic MR, Milovanovic AN, Jovic SJ, Dragin AS, Letic MDj, Miler VM. Low-level laser therapy for acute neck pain with radiculopathy: a double-blind placebo-controlled randomized study. Pain Med. 2010 Aug;11(8):1169-78. doi: 10.1111/j.1526-4637.2010.00907.x. PMID 20704667
- [Background] Ahmed I, Bandpei MAM, Gilani SA, Ahmad A, Zaidi F. Effectiveness of Low-Level Laser Therapy in Patients with Discogenic Lumbar Radiculopathy: A Double-Blind Randomized Controlled Trial. J Healthc Eng. 2022 Feb 27;2022:6437523. doi: 10.1155/2022/6437523. eCollection 2022. PMID 35265302
- [Background] Ahmed I, Mohseni Bandpei MA, Gilani SA, Ahmad A, Zaidi F. Correlation Analysis Between Pain Intensity, Functional Disability and Range of Motion Using Low-Level Laser Therapy in Patients With Discogenic Lumbar Radiculopathy: A Cross-sectional Study. J Lasers Med Sci. 2022 Jun 6;13:e26. doi: 10.34172/jlms.2022.26. eCollection 2022. PMID 36743144
- [Background] Danazumi MS, Bello B, Yakasai AM, Kaka B. Two manual therapy techniques for management of lumbar radiculopathy: a randomized clinical trial. J Osteopath Med. 2021 Feb 26;121(4):391-400. doi: 10.1515/jom-2020-0261. PMID 33705612
- [Background] Rogerson A, Aidlen J, Jenis LG. Persistent radiculopathy after surgical treatment for lumbar disc herniation: causes and treatment options. Int Orthop. 2019 Apr;43(4):969-973. doi: 10.1007/s00264-018-4246-7. Epub 2018 Nov 29. PMID 30498910
- [Background] Kostadinovic S, Milovanovic N, Jovanovic J, Tomasevic-Todorovic S. Efficacy of the lumbar stabilization and thoracic mobilization exercise program on pain intensity and functional disability reduction in chronic low back pain patients with lumbar radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(6):897-907. doi: 10.3233/BMR-201843. PMID 32675390
- [Background] Ghasabmahaleh SH, Rezasoltani Z, Dadarkhah A, Hamidipanah S, Mofrad RK, Najafi S. Spinal Manipulation for Subacute and Chronic Lumbar Radiculopathy: A Randomized Controlled Trial. Am J Med. 2021 Jan;134(1):135-141. doi: 10.1016/j.amjmed.2020.08.005. Epub 2020 Sep 13. PMID 32931763